CLINICAL TRIAL: NCT00987051
Title: Validation of the Sentinel Node in Endometrial Cancer
Brief Title: Sentinel Node and Endometrial Cancer
Acronym: Senti-Endo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P060229
Record Dates: First submitted 2009-07-30; First posted 2009-09-30 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Endometrial Neoplasms
Keywords: sentinel node procedure; radiocolloid; patent blue
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients with endometrial cancer
  Interventions: Procedure: Detection of sentinel node

INTERVENTIONS:
Procedure: Detection of sentinel node — Coelioscopy or laparotomy (based on the tumor size) after a colorimetric tracer injection

SUMMARY:
The purpose of this study is to investigate the relevance of sentinel node in endometrial cancer. Sentinel node is thought to reflect the status of lymph node. Only 10 to 20% of women with endometrial cancer exhibit lymph node metastasis hence systematic lymphadenectomy is questionable. In breast cancer, melanoma and vulvar cancer, sentinel node has emerged as an alternative to complete lymphadenectomy.

DETAILED DESCRIPTION:
To investigate the relevance of sentinel node in endometrial cancer. Sentinel node is though to reflect the status of lymph node. Only 10 to 20% of women with endometrial cancer exhibit lymph node metastasis hence systematic lymphadenectomy is questionable. In breast cancer, melanoma and vulvar cancer, sentinel node has emerged as an alternative to complete lymphadenectomy. The objective of our trial is to validate the concept of sentinel node in endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old with a surgery planned for endometrial cancer
* endometrial cancer proved by biopsy
* early stage of endometrial cancer (FIGO stage 1-2)
* without contraindication to surgery
* inform consent signed
* affiliated to general health system

Exclusion Criteria:

* endometrial cancer FIGO stages 3-4
* previous history of surgery modifying lymphatic drainage (conization myomectomy)
* pregnant women or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Detection and false negative rates of sentinel node | During the surgery (hysterectomy)

SECONDARY OUTCOMES:
Morbidity and recurrence rates | During 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Emile DARAÏ, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Tenon Hospital, Paris, France

REFERENCES:
- [Derived] Darai E, Dubernard G, Bats AS, Heitz D, Mathevet P, Marret H, Querleu D, Golfier F, Leblanc E, Rouzier R, Ballester M. Sentinel node biopsy for the management of early stage endometrial cancer: long-term results of the SENTI-ENDO study. Gynecol Oncol. 2015 Jan;136(1):54-9. doi: 10.1016/j.ygyno.2014.09.011. Epub 2014 Oct 22. PMID 25450151
- [Derived] Ballester M, Dubernard G, Lecuru F, Heitz D, Mathevet P, Marret H, Querleu D, Golfier F, Leblanc E, Rouzier R, Darai E. Detection rate and diagnostic accuracy of sentinel-node biopsy in early stage endometrial cancer: a prospective multicentre study (SENTI-ENDO). Lancet Oncol. 2011 May;12(5):469-76. doi: 10.1016/S1470-2045(11)70070-5. Epub 2011 Apr 12. PMID 21489874